CLINICAL TRIAL: NCT01671904
Title: A Phase IB, Open-Label Study Evaluating the Safety and Pharmacokinetics of Venetoclax (GDC-0199, ABT-199) in Combination With Bendamustine+Rituximab (BR) or Bendamustine+Obinutuzumab (BG) in Patients With Relapsed/Refractory or Previously Untreated Chronic Lymphocytic Leukemia
Brief Title: A Study of Venetoclax in Combination With Bendamustine + Rituximab or Bendamustine + Obinutuzumab in Participants With Relapsed/Refractory or Previously Untreated Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO28440; 2012-002351-42 (EudraCT Number)
Record Dates: First submitted 2012-08-10; First posted 2012-08-24 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; obinutuzumab; Rituximab; venetoclax

ARMS (3):
- 1L CLL BR+V (Experimental): Participants with first-line (1L)/previously untreated CLL were administered escalating doses of venetoclax (V) in combination with fixed dose bendamustine and rituximab (BR). Participants received six 28-day cycles of BR+V. Participants with 1L CLL received 6 months of single-agent venetoclax for a total of 1-year treatment duration. Single-agent venetoclax could be extended if there was detectable minimal residual disease (MRD) in the bone marrow and/or partial response (PR) after 1 year of treatment and upon the request of the treating physician.
  Interventions: Drug: Bendamustine; Drug: Rituximab; Drug: Venetoclax
- 1L CLL BG+V (Experimental): Participants with first-line (1L)/previously untreated CLL were administered escalating doses of venetoclax (V) in combination with fixed dose bendamustine and obinutuzumab (BG). Participants received six 28-day cycles of BG+V. Participants with 1L CLL received 6 months of single-agent venetoclax for a total of 1-year treatment duration. Single-agent venetoclax could be extended if there was detectable minimal residual disease (MRD) in the bone marrow and/or partial response (PR) after 1 year of treatment and upon the request of the treating physician.
  Interventions: Drug: Bendamustine; Drug: Obinutuzumab; Drug: Venetoclax
- R/R CLL BR+V (Experimental): Participants with relapsed/refractory (R/R) CLL were administered escalating doses of venetoclax (V) in combination with fixed dose bendamustine and rituximab (BR). Participants received six 28-day cycles of BR+V. Participants with R/R CLL continued single-agent venetoclax until disease progression, death, or unacceptable toxicity.
  Interventions: Drug: Bendamustine; Drug: Rituximab; Drug: Venetoclax

INTERVENTIONS:
Drug: Bendamustine — Participants will receive intravenous (IV) infusion of bendamustine (90 or 70 milligrams per square meter [mg/m^2]) on Days 2-3 of Cycle 1 and Days 1-2 of Cycles 2-6.
Drug: Obinutuzumab — Participants will receive IV infusion of obinutuzumab (100 milligrams [mg]) on Day 1 of Cycle 1; 900 mg administered on Day 2 of Cycle 1; and 1000 mg administered on Days 8 and 15 of Cycle 1 and on Day 1 of Cycles 2-6.
  Other Names: GA101; RO5072759
  Arms: 1L CLL BG+V
Drug: Rituximab — Participants will receive IV infusion of rituximab (375 mg/m^2) on Day 1 of Cycle 1 and 500 mg/m^2 administered on Day 1 of Cycles 2-6.
  Other Names: MabThera; Rituxan
  Arms: 1L CLL BR+V; R/R CLL BR+V
Drug: Venetoclax — Participants will receive multiple doses of venetoclax orally once daily.
  Other Names: ABT-199; GDC-0199

SUMMARY:
This multi-center, open-label, dose-finding study will evaluate the safety and pharmacokinetics of venetoclax (GDC-0199, ABT-199) administered in combination with bendamustine and rituximab (BR) (MabThera/Rituxan) or bendamustine and obinutuzumab (BG) to participants with first-line (1L)/previously untreated or relapsed/refractory (R/R) chronic lymphocytic leukemia (CLL). The study will explore two venetoclax combination regimens in participants with 1L CLL: BR+venetolax (V) and BG+V. Participants with R/R CLL will be administered BR+V.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing/refractory or previously untreated CLL
* Eastern Cooperative Oncology Group (ECOG) performance score of less than equal to (</=) 1
* Adequate bone marrow function
* Adequate coagulation, renal and hepatic function
* Hematological values within the limits independent of growth factor support or transfusion unless cytopenia is caused by the underlying disease, i.e., no evidence of additional bone marrow dysfunction (e.g., myelodysplastic syndrome, hypoplastic bone marrow)

Exclusion Criteria:

* Participants received an allogeneic stem cell transplant
* Known human immunodeficiency virus (HIV) positivity
* Uncontrolled autoimmune hemolytic anemia or thrombocytopenia
* Positive test results for chronic hepatitis B infection and hepatitis C virus (HCV)
* Received any anti-cancer therapy including chemotherapy or radiotherapy, steroid therapy for anti-neoplastic intent, and investigational therapy, including targeted small molecule agents within 28 days prior to the first dose of study drug or has not recovered to less than Grade 2 clinically significant adverse effect(s)/toxicity(s) of the previous therapy
* Significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, cardiovascular, or hepatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-01-13 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose Limiting Toxicities (DLTs) | Schedule (Sch) A (venetoclax [V] introduced before other agents): Cycle 1 Day 1 (Cy1D1) to Cy1D21; Sch B (V introduced after other agents): Cy1D21 to Cy2D28; Cycle length = 28 days.
  DLTs in this study were defined as specific adverse events (AEs) occurring during the DLT observation window: 1) Grade 4 neutropenia not responsive to granulocyte colony stimulating factors (G-CSF) lasting more than 14 days; 2) Grade 3 or 4 febrile neutropenia with fever lasting longer than 4 days; 3) Grade 4 thrombocytopenia resulting in bleeding, or that did not improve to Grade </=2 within 3 weeks; 4) Clinical tumor lysis syndrome (TLS) defined by the presence of laboratory TLS and one or more clinical manifestations related to the electrolyte abnormalities; 5) Grade 4 infusion-related reactions (IRRs) secondary to rituximab or obinutuzumab despite appropriate premedication and administration rate; 6) All other Grades 3, 4, or 5 AEs persisting for more than 2 weeks with or without treatment with some exceptions.

SECONDARY OUTCOMES:
Plasma Concentrations of Venetoclax | Sch A: Ramp-up D1, 8, 15, 22, 29: predose (pd), 8 h; Cy1D1: pd; Cy1D3: pd, 2, 4, 6, 8, 10 h; Cy2D1, Cy4D1, Cy6D1: pd. Sch B: Cy1D1: pd; Cy1D22, Cy2D1, Cy2D8, Cy2D15, Cy2D22 (ramp-up): pd, 8 h; Cy3D1: pd, 2, 4, 6, 8 h; Cy4D1, Cy6D1: pd.
Serum Concentrations of Rituximab | Sch A: Cy1D1, Cy2D1, Cy4D1, Cy6D1: predose, end of infusion. Sch B: Cy1D1: predose, end of infusion; Cy2D1, (ramp-up): predose, end of infusion; Cy3D1, Cy4D1, Cy6D1: predose.
Serum Concentrations of Obinutuzumab | Sch A: Cy1D1, Cy1D2: pd, end of infusion (EoI); Cy1D3: pd; Cy1D8, Cy1D15, Cy2D1: pd, EoI; Cy3D1, Cy4D1, Cy5D1, Cy6D1: pd; Sch B: Cy1D1, Cy1D2, Cy1D8, Cy1D15: pd, EoI; Cy1D22 (ramp-up): pd; Cy2D1, Cy3D1, Cy4D1, Cy5D1, Cy6D1: pd, EoI.
Plasma Concentrations of Bendamustine | Sch A: Cy1D2: predose, end of infusion. Sch B: Cy1D2, Cy3D2: predose, end of infusion.
Percentage of Participants With a Best Overall Response of Complete Response (CR) or Partial Response (PR) According to International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 Guidelines | Baseline up to approximately 5.75 years
  CR or CR with incomplete bone marrow recovery (CRi) or PR or nodular PR (nPR) was determined by the investigator according to IWCLL 2008 criteria. CR requires all of the following: Peripheral blood lymphocytes below 4x10^9/L, absence of lymphadenopathy by physical examination and computed tomography (CT) scan, No hepatomegaly or splenomegaly, Absence of disease or constitutional symptoms, Blood counts of neutrophils >1.5*10^9/L, platelets >100*10^9/L and hemoglobin >110 g/L, Bone marrow at least normocellular for age without clonal infiltrate (except for Cri). PR: two of the following features for at least 2 months: >/= 50% decrease in peripheral blood lymphocyte count from the pretreatment value, >/=50% reduction in lymphadenopathy, >/=50% reduction of liver and/or spleen enlargement, and at least one of the following blood counts: neutrophils >1.5*10^9/L, platelets >100*10^9/L and hemoglobin >110 g/L.
Duration of Response According to IWCLL 2008 Guidelines | Baseline up to approximately 5.75 years
  CR or CR with incomplete bone marrow recovery (CRi) or PR or nodular PR (nPR) was determined by the investigator according to IWCLL 2008 criteria. CR requires all of the following: Peripheral blood lymphocytes below 4x10^9/L, absence of lymphadenopathy by physical examination and computed tomography (CT) scan, No hepatomegaly or splenomegaly, Absence of disease or constitutional symptoms, Blood counts of neutrophils >1.5*10^9/L, platelets >100*10^9/L and hemoglobin >110 g/L, Bone marrow at least normocellular for age without clonal infiltrate (except for Cri). PR: two of the following features for at least 2 months: >/= 50% decrease in peripheral blood lymphocyte count from the pretreatment value, >/=50% reduction in lymphadenopathy, >/=50% reduction of liver and/or spleen enlargement, and at least one of the following blood counts: neutrophils >1.5*10^9/L, platelets >100*10^9/L and hemoglobin >110 g/L.
Percentage of Participants with CR | Baseline up to approximately 5.75 years
  CR or CR with incomplete bone marrow recovery (CRi) was determined by the investigator according to IWCLL 2008 criteria. CR requires all of the following: Peripheral blood lymphocytes below 4x10^9/L, absence of lymphadenopathy by physical examination and computed tomography (CT) scan, No hepatomegaly or splenomegaly, Absence of disease or constitutional symptoms, Blood counts of neutrophils >1.5*10^9/L, platelets >100*10^9/L and hemoglobin >110 g/L, Bone marrow at least normocellular for age without clonal infiltrate (except for Cri).
Progression-Free Survival (PFS) According to IWCLL 2008 Guidelines | Baseline up to approximately 5.75 years
  PFS was determined according to IWCLL 2008 criteria and defined as the time from randomization to the first occurrence of progressive disease (PD) or death. Disease progression was characterized by at least one of the following: 1) >/= 50% increase in the absolute number of circulating lymphocytes to at least 5*10^9/L, 2) Appearance of new palpable lymph nodes (> 15 mm in longest diameter) or any new extra-nodal lesion; 3) >/= 50% increase in the longest diameter of any previous site of lymphadenopathy; 4) >/= 50% increase in the enlargement of the liver and/or spleen; 5) Transformation to a more aggressive histology.
Overall Survival (OS) | Baseline up to approximately 5.75 years
  OS was defined as the time from randomization to death from any cause.
Number of Participants With Adverse Events | Up to approximately 5.75 years
  An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (12):
- United States (4):
  - University of California San Diego Medical Center, La Jolla, California
  - Ingalls Hospital; Cancer Clinical Trials, Harvey, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - North Star Lodge, Yakima, Washington
- France (4):
  - Hopital Claude Huriez, Lille
  - Hopital Saint Eloi, Montpellier
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
- Germany (4):
  - Universitatsklinik Koln, Cologne
  - Apotheke des Universitätsklinikums Freiburg, Freiburg im Breisgau
  - Klinikum Schwabing, München
  - Universtitätsklinikum Ulm; Klinik für Innere Medizin III, Ulm